CLINICAL TRIAL: NCT02083263
Title: Study of Non Invasive Ventilation With High Pressure as Airways Clearance Technique in Adults Patients With Cystic Fibrosis
Brief Title: Non Invasive Ventilation as Airway Clearance in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Cecilia Rodriguez, Specialist Physiotherapist, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF2012-1
Record Dates: First submitted 2012-11-16; First posted 2014-03-11 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Cystic Fibrosis
Keywords: Lung function
MeSH Terms: conditions — Cystic Fibrosis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilevel (Experimental): Bilevel, 3 months. The treatment was performed twice a day, 1 hour each treatment.
  Interventions: Device: Bilevel
- PEP mask (Active Comparator): PEP mask, 3 months. The treatment was performed twice a day, 1 hour each treatment.
  Interventions: Device: PEP mask

INTERVENTIONS:
Device: Bilevel — 3 months
  Arms: Bilevel
Device: PEP mask — 3 months
  Arms: PEP mask

SUMMARY:
With the use of Non invasive ventilation the patients with cystic fibrosis will have better lung function (FEV1).

DETAILED DESCRIPTION:
3 months intervention between PEP an Bilevel. The patients will follow up under 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF older than 18 years
* FEV1 between 20% and 69% of predictive.
* No acute exacerbation.
* No Burkhordelia Cepacia/MRSA colonization.

Exclusion Criteria:

* Children under 18 year
* acute exacerbation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Rodriguez, Physio, Principal Investigator — Karolinska Institutet
Locations (1):
- Cecilia Rodriguez, Stockholm, Stockholm County, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilevel: Bilevel, 3 months
  Bilevel: 3 months
- PEP Mask: PEP mask, 3 months
  PEP mask: 3 months
Period: Overall Study
Arm/Group | Bilevel | PEP Mask
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilevel | PEP Mask | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (11) | 33 (9) | 31 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Sweden | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Lung Function: Lung Clearance Index
Description: Lung clearance index was calculated as the number of lung volume turnovers (cumulative expired volume divided by the functional residual capacity) required to reduce end-tidal nitrogen concentration to 1/40th of the starting value.
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: lung clearance index
Arm/Group | Bilevel | PEP Mask
Number analyzed (Participants) | 16 | 16
lung clearance index | 9 (3) | 9.7 (3)

2. Secondary Outcome: Blood Gases:1 Month After Chest Physiotherapy Will Take Blood Gases (Kpa).
Description: After physiotherapy will take blood gases (kpa) before chest physiotherapy and perform once a month.
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bilevel | PEP Mask
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes